CLINICAL TRIAL: NCT01019460
Title: A Comparative Study of Capsule Endoscopy, Magnetic Resonance Imaging and Computer Tomography Scanning of the Small Bowel in Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Michael Dam Jensen, Dr, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: S-20070072
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Crohn's Disease
Keywords: Small intestine; Magnetic resonance imaging; Computed tomography scanning; Capsule endoscopy
MeSH Terms: conditions — Crohn Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Magnetic resonance imaging, computed tomography scanning and capsule endoscopy — All patients are examined with ileo-colonoscopy, capsule endoscopy, MRI and CT of the small bowel within 14 days. Capsule endoscopy will not be performed in patients with small bowel stenosis confirmed at ileo-colonoscopy, MRI and/or CT.

SUMMARY:
The aim of this study is to evaluate three diagnostic methods for assessing small bowel disease in patients with suspected or known Crohn's disease. All patients are examined with ileo-colonoscopy, capsule endoscopy, MRI and CT of the small bowel within 14 days. However, capsule endoscopy is not performed in patients with stenosis detected at ileo-colonoscopy, MRI and/or CT. All investigations are described in a similar pre-defined and standardized fashion and the radiologist and physician responsible for describing the findings at MRI, CT and capsule endoscopy are blinded to the findings at ileo-colonoscopy. The physician in charge of treatment receives a randomised result of either MRI, CT or capsule endoscopy. Thereafter patients are followed during 12 months to evaluate differences in clinical outcome depending on the randomized result. In combination with the diagnostic validity and inter-observer agreement of MRI, CT and capsule endoscopy we seek to establish the optimal diagnostic strategy in these two patient categories.

DETAILED DESCRIPTION:
OVERALL AIM OF THE STUDY To evaluate three diagnostic methods for assessment of intestinal disease in patients with suspected or newly diagnosed Crohn's disease and patients with known Crohn's disease.

PARTICIPATING CENTRES

* Department of Medical Gastroenterology, Odense University Hospital, DK-5000 Odense C
* Department of Internal Medicine, section of Gastroenterology, Vejle Hospital, DK-7100 Vejle
* Department of Internal Medicine, section of Gastroenterology, Sydvestjysk Hospital, DK-6700 Esbjerg
* Department of Internal Medicine, section of Gastroenterology, Svendborg Hospital, DK-5700 Svendborg
* Department of Radiology, Vejle Hospital, DK-7100 Vejle

PROTOCOL A

A comparative study of capsule endoscopy, magnetic resonance imaging and computer tomography scanning of the small bowel in patients with suspected or newly diagnosed Crohn's disease

Protocol procedures:

At inclusion all patients will have a standardised work-up including medical history, physical examination, blood and faeces samples and ileo-colonoscopy. Within two weeks MRI and CT scanning of the small intestine (on the same day and in randomised order) and subsequently CE will be performed in all patients. All investigations are described in a similar pre-defined and standardized fashion and the radiologist and physician responsible for describing the findings at MRI, CT and CE are blinded to the findings at ileo-colonoscopy and the other small bowel examinations. In the follow-up part of the study the physician in charge of the patient will be randomised to receive the results of either MRI, CT or CE.

Anticipated outcome:

The study is performed to improve evidence about what is the best primary investigation for assessment of small intestinal involvement in patients with suspected Crohn's disease, to evaluate if a combination of diagnostic modalities may improve our assessment of disease burden for the individual patients, to study whether the initial diagnostic modalities affect the handling of the patients and to study the interobserver variation of MRI and CT scanning.

PROTOCOL B

A comparative study of magnetic resonance imaging, computer tomography scanning and capsule endoscopy in patients with known Crohn's disease

Protocol procedures:

At inclusion all patients will undergo a standardised work-up including history, physical examination, blood and faeces samples and ileo-colonoscopy. Within two weeks MRI, CT scanning of the small intestine (on the same day in randomised order) and capsule endoscopy will be performed in all patients. Capsule endoscopy will not be performed in patients with small bowel stenosis confirmed at ileo-colonoscopy, MRI and/or CT. All three investigations will be described in a similar predefined standardized fashion with the radiologist blinded to the findings at ileo-colonoscopy. In the randomised part of the study the physician in charge of the patient will be randomised to receive the result of either MRI, CT og capsule endoscopy.

Anticipated outcome:

The best diagnostic method for evaluation of small intestinal involvement in patients with known Crohn's disease may be different from patients suspected of Crohn's disease. Thus in the current study we hope to provide evidence of whether MRI, CT scanning or capsule endoscopy is the best diagnostic approach.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Age > 15 years
* Written informed consent

Patients with established CD are included if assessment of small bowel disease was necessary prior to expected surgery or a change in medical therapy.

Patients with suspected CD are included on either clinical, endoscopical or histological criteria or a combination of these.

* Clinical criteria: Diarrhoea and/or abdominal pain for more than 1 month (or repeated episodes of diarrhoea and/or abdominal pain) associated with one or more of the following findings: CRP > 5 mg/l, thrombocytosis, anaemia, fever, weight loss, perianal abscess/fistula or a family history of inflammatory bowel disease.
* Endoscopical criteria (at least one): Ulcerations and/or stenosis in the terminal ileum, inflammation in the colon not involving the rectum, and aphthous ulcerations in the colon.
* Histological criteria (at least one): Epitheloid cell granulomas, chronic inflammation in the lamina muscularis mucosae or deeper and chronic inflammation in the colon not involving the rectum.

Exclusion Criteria:

* Acute bowel obstruction, elevated serum-creatinine, severe claustrophobia, cardiac pacemaker, implanted magnetic foreign bodies, use of NSAID's, pregnancy and lactation

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for CT scanning of the small bowel, MRI of the small bowel and CE. | February 2010

SECONDARY OUTCOMES:
Interobserver variation for capsule endoscopy, MRI and CT scanning of the small intestine Patient experienced discomfort | February 2010

REFERENCES:
- [Derived] Jensen MD, Andersen RF, Christensen H, Nathan T, Kjeldsen J, Madsen JS. Circulating microRNAs as biomarkers of adult Crohn's disease. Eur J Gastroenterol Hepatol. 2015 Sep;27(9):1038-44. doi: 10.1097/MEG.0000000000000430. PMID 26230660
- [Derived] Jensen MD, Nathan T, Rafaelsen SR, Kjeldsen J. Ileoscopy reduces the need for small bowel imaging in suspected Crohn's disease. Dan Med J. 2012 Sep;59(9):A4491. PMID 22951194